CLINICAL TRIAL: NCT00544193
Title: Pilot Study of Gemcitabine and IORT/EBRT in Locally Advanced Upper Gastrointestinal Malignancies
Brief Title: Gemcitabine and Radiation Therapy in Treating Patients With Locally Advanced Upper Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 97087; P30CA033572 (NIH); CHNMC-97087
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the gallbladder; adenocarcinoma of the pancreas; adenocarcinoma of the stomach; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; localized extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; localized gallbladder cancer; recurrent gallbladder cancer; unresectable gallbladder cancer; recurrent gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; stage I gastric cancer; recurrent pancreatic cancer; small intestine adenocarcinoma; stage IV pancreatic cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms | interventions — Gemcitabine; Polymerase Chain Reaction; Immunohistochemistry; Radiotherapy

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Genetic: polymerase chain reaction
Other: immunohistochemistry staining method
Procedure: conventional surgery
Radiation: intraoperative radiation therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gemcitabine when given together with radiation therapy in treating patients with locally advanced upper gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the feasibility of combining preoperative or intraoperative gemcitabine hydrochloride with intraoperative radiotherapy.
* To determine the tolerance of gemcitabine hydrochloride given concurrently with external-beam radiotherapy.
* To measure biochemical parameters in tumors that may correlate with the effectiveness of therapy.

OUTLINE: Patients receive gemcitabine hydrochloride IV 12-18 hours prior to planned surgery. All patients then undergo an exploratory laparotomy that may include tumor debulking, Whipple-type resection (pancreaticoduodenectomy), total pancreatectomy, gastrojejunostomy, total or partial gastrectomy, or cholecystectomy and en bloc resection depending on the extent of the disease. Patients with no metastatic disease beyond regional lymph nodes also undergo intraoperative radiotherapy.

Beginning 2-6 weeks after surgery, patients undergo external-beam radiotherapy (EBRT) once a day 5 days a week for up to 7 weeks. Patients also receive escalating doses of gemcitabine hydrochloride IV at the beginning of each week of EBRT.

Patients undergo tissue sample collection periodically for correlative studies. Samples are analyzed for thymidylate synthase (TS), ribonucleotide reductase (RR), excision-repair-cross-complementing (ERCC)-1 protein, deoxycytidine kinase mRNA. Biopsy tissues are also analyzed for gemcitabine triphosphate, dATP, and dCTP content. p53 status is assessed via immunohistochemistry and mRNA levels via quantitative polymerase chain reaction (PCR).

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then once a year thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following upper gastrointestinal malignancies:

  * Localized pancreatic adenocarcinoma

    * Stage I, II, or III disease
    * Parapancreatic node involvement and locally recurrent disease allowed
  * Locally advanced biliary, gallbladder, or ampullary adenocarcinoma

    * Stage II, III, or locally recurrent disease
  * Histologically confirmed locally advanced gastric adenocarcinoma

    * T3, T4, or node positive OR locally recurrent disease
  * Histologically confirmed locally advanced duodenal cancer

    * Stage II or III disease
* Locally advanced, but unresectable cancers may be included on protocol if appropriate for intraoperative radiotherapy (IORT)
* Other histologies may be considered for this protocol except for lymphoma, sarcoma, or neuroendocrine tumors
* Patients with evidence of metastatic disease are eligible if there is significant local disease warranting surgery and IORT

PATIENT CHARACTERISTICS:

* Karnofsky performance status > 60%
* Life expectancy > 4 months
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Serum creatinine < 2.0 mg/dL
* ALT < 3 x normal
* Bilirubin < 2 x normal
* Must be able to give voluntary informed consent
* No severe intercurrent illness that would make the patient inappropriate for laparotomy or otherwise inappropriate for treatment on protocol
* Prior history of malignancy allowed

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin C)
* Prior gemcitabine hydrochloride allowed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1997-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Feasibility
Tolerance
Measurement of biochemical parameters in tumors that may correlate with the effectiveness of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I. Shibata, MD, Study Chair — City of Hope Comprehensive Cancer Center